# **Clinical Trial Protocol**

#### Title

Effectiveness of Gait Retraining in Female Runners with Patellofemoral Pain: A Randomized Controlled Trial

#### 1. Administrative Information

Sponsor / Responsible Party: Beijing Sport University

Collaborators: Sports Medicine Center, West China Hospital, Sichuan University

Principal Investigator: Haonan Wang, PhD

Trial Registration: ClinicalTrials.gov (to be assigned)

Ethics Approval: Approved by Ethics Committee of Beijing Sport University

Study Period: December 2022 - December 2023

## 2. Background and Rationale

Patellofemoral pain (PFP) is the most common running-related overuse injury, with prevalence up to 17% among runners. Increased patellofemoral joint stress (PFJS) is a major biomechanical contributor to PFP. Traditional strengthening exercises improve function but do not alter running biomechanics. Gait retraining, particularly cadence modification, has been proposed as a promising approach to reduce PFJS and alleviate symptoms. However, evidence from randomized controlled trials remains limited. This study investigates whether wearable device-assisted gait retraining reduces pain, improves function, and modifies running biomechanics in female runners with PFP compared to education alone.

# 3. Objectives

Primary Objective: To determine the effectiveness of wearable device-assisted gait retraining on pain reduction during running in female runners with PFP.

## Secondary Objectives:

- To assess improvements in function (Anterior Knee Pain Scale, AKPS)
- To examine changes in running mechanics (knee kinematics, kinetics, PFJS)
- To evaluate adherence, feasibility, and safety of wearable device-assisted gait retraining

## 4. Study Design

Type: Randomized, controlled, single-blind, parallel-group trial

Allocation: 1:1 randomization

Masking: Outcome assessors blinded; participants not blinded due to intervention nature Arms:

- Intervention Arm: Education + Wearable device-assisted gait retraining
- Control Arm: Education only

Study Duration: 18 weeks per participant (6-week intervention + 12-week follow-up)

# 5. Participants

**Inclusion Criteria:** 

- Female, age 18-45 years
- Unilateral/bilateral anterior knee pain > 4 weeks
- VAS pain  $\geq 3/10$  during running and  $\geq 2$  of the following: jumping, squatting, kneeling, stairs, prolonged sitting, or resisted knee extension
- Running ≥ 15 km per week
- Natural rearfoot striker (verified by high-speed video)

**Exclusion Criteria:** 

- Acute trauma, history of patellar dislocation, meniscal/chondral lesions
- Prior knee surgery or injection in past 12 months
- Rheumatologic, neurologic, or degenerative disease

- Pregnancy

#### 6. Interventions

## **6.1 Control Group (Education)**

Delivered via WeChat platform. Content: PFP education, load management strategies, symptom-based training modifications, and strengthening exercises (quadriceps & hip). Self-monitored running program guided by pain thresholds.

#### **6.2 Intervention Group (Gait Retraining + Education)**

Same education program as control. Gait retraining protocol: 6-week program, twice per week. Step rate increased by 10%, monitored via smartwatch (Huawei GT4). Real-time cadence feedback via auditory metronome cues. Feedback frequency: every session (weeks 1–4), once (week 5), faded (week 6). Duration progressed from 15 min to 30 min per session. Pain monitoring:  $\leq 3/10$  during running, return to baseline within 60 min.

#### 7. Outcomes

#### **7.1 Primary Outcome**

Pain during running (VAS-R, 0–100 mm) at baseline, 6 weeks, and 18 weeks

## **7.2 Secondary Outcomes**

- VAS-U (usual pain), VAS-W (worst pain)
- Function: Anterior Knee Pain Scale (AKPS)
- Running-related measures: weekly mileage, cadence (smartwatch logs)
- Running mechanics: 3D kinematics, GRF, PFJS and contact force calculations

#### **7.3 Safety Outcomes**

Adverse events (pain exacerbation, injuries, withdrawal)

## 8. Sample Size

Sample size estimated with G\*Power. Detectable difference: 20 mm VAS (MCID for PFP). Power: 80%,  $\alpha$  = 0.05. Estimated: 22 participants per group (total n=44), accounting for 15% dropout.

## 9. Randomization and Blinding

Random sequence generated by independent statistician. Allocation concealed in sequential opaque envelopes. Assessors blinded to group assignment. Participants instructed not to disclose intervention to evaluators.

# 10. Data Analysis

Approach: Intention-to-treat and per-protocol. Statistical tests: Repeated measures ANOVA and linear regression models (adjusted for baseline, age, BMI, running duration, symptom duration). Multiple imputation for missing data. Effect size: Partial eta squared ( $\eta^2$ ). Significance: p < 0.05.

#### 11. Ethics and Dissemination

Ethical approval granted by Beijing Sport University Ethics Committee. Informed consent obtained from all participants. Results will be disseminated via peer-reviewed journals, academic conferences, and ClinicalTrials.gov.